CLINICAL TRIAL: NCT02482168
Title: Phase 1 Study to Evaluate the Safety and Tolerability of the CD40 Agonistic Monoclonal Antibody APX005M in Subjects With Solid Tumors
Brief Title: Study of the CD40 Agonistic Monoclonal Antibody APX005M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apexigen America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APX005M-001
Record Dates: First submitted 2015-06-11; First posted 2015-06-26 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cancer; NSCLC; Melanoma; Urothelial Carcinoma; MSI-H; Head and Neck Cancer
Keywords: immunotherapy; CD40
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Transitional Cell; Head and Neck Neoplasms | interventions — sotigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- APX005M every 3 week (Experimental): Subjects receive APX005M intravenously every 3 week until disease progression, unacceptable toxicity or death.
  Interventions: Drug: APX005M
- APX005M every 2 week (Experimental): Subjects receive APX005M intravenously every 2 week until disease progression, unacceptable toxicity or death.
  Interventions: Drug: APX005M
- APX005M every 1 week (Experimental): Subjects receive APX005M intravenously every 1 week until disease progression, unacceptable toxicity or death.
  Interventions: Drug: APX005M

INTERVENTIONS:
Drug: APX005M — APX005M is a CD40 agonistic monoclonal antibody

SUMMARY:
This study is a phase 1 open-label dose escalation study of the immuno-activating monoclonal antibody APX005M in adults with solid tumors. Study is intended to establish the maximum tolerated dose and the overall safety and tolerability of APX005M in 3 different administration schedules.

DETAILED DESCRIPTION:
APX005M-001 is an open-label study and comprises a dose-escalation portion of approximately 8 dose level cohorts, plus an expansion cohort.

Eligible subjects with solid tumors will receive intravenous APX005M every 3 week, every 2 week or every 1 week until disease progression, unacceptable toxicity or death, whichever occurs first.

Study objectives include:

* Evaluate safety of APX005M
* Determine the maximum tolerated dose of APX005M
* Determine the pharmacokinetic parameters of APX005M: the maximal drug concentration (Cmax), area under the curve of serum concentration over time (Area Under the Curve/ AUC), and half-life (t½).
* Preliminary assessment of clinical response

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically documented diagnosis of solid tumor
* For subjects in the every 2 week and every 1 week dosing cohorts histologically or cytologically documented diagnosis of urothelial carcinoma, melanoma, squamous cell carcinoma of the head and neck, non-small cell lung cancer, or any solid tumor with high microsatellite instability status (MSI-high)
* No known effective therapy options are available
* Measurable disease by RECIST 1.1
* ECOG performance status of 0 or 1
* Adequate bone marrow, liver and kidney function
* No toxicities related to prior treatment related toxicities with the exception of alopecia and neuropathy
* Negative pregnancy test for women of child bearing potential

Key Exclusion Criteria:

* Any history of or current hematologic malignancy
* Major surgery or treatment with any other investigational agent within 4 weeks
* Uncontrolled diabetes or hypertension
* History of arterial thromboembolic event
* History of congestive heart failure, symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction
* Active known clinically serious infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 28 days following first dose of APX005M
  The rate of DLTs will be assessed in approximately 56 subjects. DLTs will include Grade 4 neutropenia, anemia, thrombocytopenia, Grade 3or 4 nausea, cytokine release syndrome and other Grade 3 non-hematological toxicity
Incidence of adverse events | Through up to approximately 4 weeks following last dose of APX005M
  Incidence and severity of AEs and specific laboratory abnormalities graded according to NCI-CTCAE, v4.03

SECONDARY OUTCOMES:
Blood concentrations of APX005M | Predose, 0.5, 1, 2, 4, 24, 48 and 168 hours following first and third dose of APX005M
  PK parameters of APX005M
Presence and titer of anti-APX005M antibodies | Prior to first dose, approximately 3, 6 and 9 weeks following first dose and approximately 4 weeks following last dose of APX005M
  Assess incidence of anti-drug antibodies (ADA)
Objective response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) | Every 8 weeks up to approximately 1 year following first dose of APX005M
  Efficacy assessments will follow RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Apexigen America, Inc.
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Case Western Reserve University, Cleveland, Ohio
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania